CLINICAL TRIAL: NCT04583124
Title: Neurotoxicity Prevention With a Multimodal Program (ATENTO) Prior to Cancer Treatment Versus Throughout Cancer Treatment in Women Newly Diagnosed for Breast Cancer: a Randomized Clinical Trial.
Brief Title: Adjusting the Dose of Therapeutic Exercise to Prevent Neurotoxicity Due to Anticancer Treatment (ATENTO)
Acronym: ATENTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Asociación Española contra el Cáncer (Other)
Responsible Party: Principal Investigator, Irene Cantarero Villanueva, Irene Cantarero Villanueva, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATENTO19
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasm
Keywords: Breast neoplasm; Breast cancer; Therapeutic Exercise; Neurotoxicity; Vagal activation techniques
MeSH Terms: conditions — Breast Neoplasms; Neurotoxicity Syndromes | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATENTO-B (Experimental): A multimodal program based on adapted therapeutic exercise and vagal activation techniques performed before the begining of medical treatment for breast cancer. It consits of 18 sessions to perform aerobic and strength exercises (90' approximately plus myofascial stretching and breathing exercises (20'). Frequency of sessions will be adapted to the recovery of each patients (by heart rate variability parameters and patient perception).
  ATENTO is divided in two parts: a) general phase: aimed to improve the overall physical health condition and to correctly learn the execution of each exercise (2 weeks); and b) specific phase: aimed to neurotoxicity prevention.
  Interventions: Other: ATENTO-B
- ATENTO-T (Active Comparator): A multimodal program based on adapted therapeutic exercise and vagal activation techniques performed throughout medical treatment for breast cancer. It consits of 18 sessions to perform aerobic and strength exercises (90' approximately plus myofascial stretching and breathing exercises (20'). Frequency of sessions will be adapted to the recovery of each patients (by heart rate variability parameters and patient perception).
  ATENTO is divided in two parts: a) general phase: aimed to improve the overall physical health condition and to correctly learn the execution of each exercise (2 weeks); and b) specific phase: aimed to neurotoxicity prevention.
  Interventions: Other: ATENTO-T

INTERVENTIONS:
Other: ATENTO-B — Patients will perform therapeutic exercise and vagal activation techniques before medical treatment and will follow the usual care after medical treatment.
  Other Names: Multimodal program (therapeutic exercise and vagal activation techniques) before medical treatment
  Arms: ATENTO-B
Other: ATENTO-T — Patients will perform therapeutic exercise and vagal activation techniques throughout medical treatment and will follow the usual care after medical treatment.
  Other Names: Multimodal program (therapeutic exercise and vagal activation techniques) throughout medical treatment
  Arms: ATENTO-T

SUMMARY:
The purpose of this study is to determine whether a multimodal program based on therapeutic exercise and vagal activation techniques for newly diagnosed breast cancer women has better results in terms of neurotoxicity prevenion before or during medical treatments.

DETAILED DESCRIPTION:
One of the most common side effects of breast cancer and its treatments is neurotoxicity of central and peripheral nervous system. Neurotoxicity is present in up to 75% of this population, which implies a large impact in quality of life. There is a special interest in the preventive possibilities of therapeutic exercise relating to these neurological sequelae, whose benefits could improve thanks to the combination with vagal activation techniques.

This superiority randomized controlled trial will be aimed to check the effects of a multimodal intervention (ATENTO) based on moderate-high intensity and individualized therapeutic exercise (aerobic and strength exercises) and vagal activation techniques (myofascial stretching and breathing exercises), on neurotoxicity prevention in women with breast cancer before starting potentially neurotoxic treatments (ATENTO-B) versus throughout them (ATENTO-T). A sample of 56 women newly diagnosed with breast cancer calculated with a power of 85% will be allocated into two groups.

This study could provide an impetus for the introduction of early multimodal intervention methods of preventing neurotoxicity and consequently avoid the current QoL deterioration that breast cancer patients suffer throughout their treatments.

ELIGIBILITY:
Inclusion Criteria:

* To have 18 years or older
* To have a breast cancer diagnosis (Stage I-III)
* To be on waiting list for medical adjuvant treatment with risk of central and/or peripheral neurotoxicity.
* To have signed the informed consent.
* To have medical clearance for participation.

Exclusion Criteria:

* To have a previous history of cancer or any cancer treatment.
* Pregnant patients.
* To participate in another intervention that could influence on the outcomes.
* To have a neurodegenerative disease that affects central or peripheral nervous system and could influence the results.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Quality of life (QLQ) | Participants will be followed over 12 months
  The primary outcome will be assessed with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0, that is one of the most widely used instruments to measure quality of life in cancer patients.

SECONDARY OUTCOMES:
Cognitive function: attention | Participants will be followed over 12 months
  The Trail Making Test will be used to assess speed for attention, sequencing, mental flexibility, visual search and motion function.
Cognitive function: memory and processing speed | Participants will be followed over 12 months
  Wechsler Adult Intelligence Scale (WAIS-IV) will be used to assess working memory and processing speed
Subjective cognitive function | Participants will be followed over 12 months
  The Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) will be used to assess the subjective cognitive functioning.
Intensity of symptoms | Participants will be followed over 12 months
  The EORTC QLQ-Chemotherapy-induced peripheral neuropathy (QLQ-CIPN20) will be used to assess neuropathic symptoms.
Tactile sensation | Participants will be followed over 12 months
  The Semmes-Weinstein monofilaments (SWMs) will be used to detect peripheral sensory neuropathy.
Psychological diistress | Participants will be followed over 12 months
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess levels of anxiety and depression.
Presence of pain | Participants will be followed over 12 months.
  Pressure pain thresholds (PPT) will be used to explore bilaterally the quadriceps, deltoid, trapezius and cervical muscles using an algometer.
Sleep disturbance | Participants will be followed over 12 months
  The Pittsburgh Sleep Quality Index (PSQI) will evaluate the quality of sleep through seven dimensions (quality, latency, duration, efficiency, alterations, use of medication and daily dysfunction).
Cardiorespiratory fitness | Participants will be followed over 12 months
  Cardiopulmonary exercise test will be performed with a Medisoft, 870 A treadmill and Jaeger MasterScreen® CPX gas analyser to assess VO2 peak following the University of Northern Colorado Cancer Rehabilitation Institute (UNCCRI).
Static body balance | Participants will be followed over 12 months
  Flamingo test will be used to assess static body balance

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain